CLINICAL TRIAL: NCT03154788
Title: Developing and Evaluating a Series of Falls Risk Awareness Corporate Videos Which Target Community-dwelling Older People: a Sequential Mixed-method Study.
Brief Title: Falls Risk Awareness Video Study
Status: Completed | Type: Observational
Sponsor: Curtin University (Other)
Responsible Party: Principal Investigator, Lex de Jong, Research Fellow, Curtin University
Other Study IDs: HRE2017-0038
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Age Problem
Keywords: Falls prevention; Community-Based Participatory Research

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this study is to develop and evaluate three short corporate falls risk awareness videos of approximately 1-2 minutes (each) by using the feedback from community-dwelling people aged 50 years and above. The three videos aim to make a broad audience aware of the risk of falling as one gets older.

DETAILED DESCRIPTION:
Every year one in three people aged 60 years and above fall over. More than 96.000 Australians are admitted to hospital each year due to a fall and this number is rising by 2% each year. People who have had a fall account for almost 40% of all hospitalised injury cases, with almost half of those falls resulting in injuries such as broken hips, neck- and head injuries. In 2015 almost 2300 Australians died as a direct result of a fall, a number which is more than three times higher than the number of people who die in car accidents.

Given the high risk of experiencing (an) (injurious) fall(s), various campaigns have been conducted with the aim of making older people aware that it is important to prevent falls. Also, numerous resources (websites, leaflets) are available to the general public that inform them of the several activities they can undertake to reduce their risk of falls. However, these campaigns and available resources do not seem to be compelling enough. Research has shown that people over the age of 60 still tend to underestimate their own risk of a fall, and have low levels of knowledge about how to prevent falls. Also, many older people report that they are not motivated to take action to reduce their risk of falls even thought they think that falls prevention would be useful for other older people. In particular older people state that they seek out information only after they fall and not before. It would be beneficial if the broad population and people over the age of 60 in particular, were more aware about falls and more motivated to take action(s) to reduce their risk of falling. Therefore the investigators aim to develop three short falls risk awareness videos that are appealing to people of all age groups and especially people aged 60 years and above.

Based on research findings by the investigators, to date three prototype versions of short falls risk awareness videos have been developed. During this research project these videos will be evaluated and then amended and developed further according to the feedback given by the participants. The feedback from participants will be sought in two phases.

Phase 1 In the first phase 50 community-dwelling older people over the age of 50 will be invited to share their thoughts and opinions about the prototype versions of the three falls risk awareness videos. For the participants in this phase of the study it will involve attending a focus group meeting of about 1½ hour in total together with 8-10 other participants. During this focus group meeting (but prior to the actual discussion about the videos) the researchers will also ask the participants to help test a questionnaire which is developed specifically for the purpose of this study. Participants will be asked to fill in the questionnaire twice (with a 20 minute rest in between). Questions pertain to the participants' knowledge of falls and their capabilities and motivation towards undertaking fall prevention activities. The researchers plan to use this questionnaire in the second phase of the project. It this phase it is solely used to measure the time taken to complete the questionnaire and to establish its reliability (and not to actually measure the outcomes at this point). Then the prototype videos will be shown twice, followed by a discussion group of around 45-50 minutes in which several questions will be asked about the content and the appeal of the three videos. Subsequent to the focus groups, the participants' feedback on the prototype videos will be evaluated and used to amend/develop the videos further.

Phase 2 During the second phase of this research study the amended videos will be screened to a larger audience of about 100 community-dwelling people aged 50 years and above during a World Café forum. This is a research design that specifically aims to gain consumers opinions about topics of interest. The aim of this forum is to seek these people's feedback on the three videos. In addition, the researchers will evaluate if having watched these three videos has changed the forum attendees' knowledge, intentions and some basic beliefs towards falls and engaging in falls prevention activities. This will be measured using the questionnaire that was pretested for reliability in the first phase of the study. The participants' feedback about the videos will be evaluated and used to develop the final versions of the videos. These final videos will be used in a future research study, most likely by being placed online and evaluated using the questionnaire previously developed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years and older living in the (Greater) Perth region, Western Australia.
* Living independently (this can include living with others, receiving assistance for daily tasks, or living in a retirement village).
* Sufficiently mobile to attend a community focus group or World Cafe Forum (i.e. be able to leave their home with or without assistance).
* Sufficient English language skills (self-assessed) to be able to successfully join in the focus group and World Cafe forum discussion(s).
* Able to provide written informed consent.

Exclusion Criteria:

* Living in a nursing home.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Community-dwelling older people.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
Reactions to prototype versions of the three short corporate falls risk awareness videos. | 6 months.
  Qualitative data collected during focus groups (phase 1)
Reactions to prototype versions of the three short corporate falls risk awareness videos. | 18 months.
  Qualitative data collected during a World Cafe Forum (phase 2)

CONTACTS AND LOCATIONS:
Overall Officials: Lex de Jong, PhD, Principal Investigator — Curtin University
Locations (1):
- Curtin University, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Jong LD, Francis-Coad J, Wortham C, Haines TP, Skelton DA, Weselman T, Hill AM. Evaluating audio-visual falls prevention messages with community-dwelling older people using a World Cafe forum approach. BMC Geriatr. 2019 Dec 9;19(1):345. doi: 10.1186/s12877-019-1344-3. PMID 31818252